CLINICAL TRIAL: NCT01086202
Title: Clinical Outcome Comparison Between Medial and Lateral Offset Reverse Shoulder Arthroplasty
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Wesley P. Phipatanakul, M.D. Asscoaite Professor, Loma Linda University
Other Study IDs: 59247
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2011-06

CONDITIONS: Rotator Cuff Tear; Proximal Humerus Fractures; Malunions; Chronic Proximal Humerus Dislocations
Keywords: irreparable rotator cuff tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Tornier Reversed Shoulder Arthroplasty Medial Offset
- Lateral offset arthroplasty

SUMMARY:
The purpose of this study is to prospectively evaluate two FDA approved implant designs for the Tornier Reverse Shoulder arthroplasty. The small difference in design is the amount of offset each implant has. This offset may improve clinical outcomes in the patient population. There have been no clinical comparative studies between these two designs in the literature to date. We would like to follow these patients for two years after implantation of the reverse shoulder and evaluate their radiographs, pain scores, and shoulder functional scores. this would be the first randomized prospective single blinded study of its kind.

DETAILED DESCRIPTION:
The combination of shoulder arthritis and rotator cuff deficiency presents quite a surgical challenge. The reverse prosthesis offers a treatment option for subset of patients as previous attempts to treat with soft tissue reconstruction or conventional arthroplasty have provided sub-optimal clinical results. Numerous reports in the literature have validated the effectiveness of the reverse design.

Patients meeting criteria must be between the ages of 50 and 95 years of age and are a candidate for a reverse shoulder arthroplasty. This is includes patients with rotator cuff tear arthroplasty, irreparable rotator cuff tears, significant proximal humerus fractures and malunions, and chronic proximal humerus dislocators. A total of 40 patients will be enrolled and randomized to either one of two groups; 20 patients will be randomized to the Tornier Reversed shoulder Arthroplasty Medial offset, and 20 will receive the Lateral offset design. Both implants are FDA approved. The patients will be followed for 24 months and will follow-up will be at 6 weeks, 3 months, 6 months, 12 months and 24 months questionnaires will be completed at each visit, x-rays will be done at pre-op, 3 month, 6 months 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient that is a candidate for reverse shoulder arthroplasty this includes:

* rotator cuff tear arthroplasty,
* irreparable rotator cuff tear,
* significant proximal humerus fracture and malunions,
* chronic proximal humerus dislocation.

Exclusion Criteria:

1. Any patient with previous arthroplasty on affected shoulder.
2. Patient who will need additional procedures including: bone grafting of the glenoid and muscle transfer.
3. Patients who do not want to participate or participate in follow-ups.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly/aged, Inpatient and outpatient, healthy patients, females, males physically handicapped, Seventh-day Adventist cohort.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2010-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome Comparison Between Medical Lateral Offset Reverse Shoulder Arthroplasty | 36 Months
  We would like to follow these patients for two years after implantation of the reverse shoulder and evaluate their radiographs, pain scores, and shoulder functional scores. this would be the first randomized prospective single blinded study of its kind.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Phipatanakul, MD, Principal Investigator — Loma Linda University Health Dept. Orthopaedic Surgery
Locations (1):
- Loma Linda University Health Care Dept. of Orthopaedic Surgery, Loma Linda, California, United States